CLINICAL TRIAL: NCT04836793
Title: Study of Humoral and Cellular Immune Responses Following SARS-CoV-2 Vaccination to Predict Immune Responses in Cancer Patients
Brief Title: COVID-19-Study of Immune Responses Following Vaccination Against SARS-CoV-2
Acronym: CACOV-VAC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-A00166-35
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Cancer; Elderly; Healthy Aging
Keywords: vaccination; T cell; SARS-COV-2; COVID-19; cancer
MeSH Terms: conditions — Neoplasms; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — PBMC PLASMA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with cancer: * Patients with active treatment in adjuvant/induction setting,
  * Patients with active treatment in metastatic/relapse setting,
  * Patients without active treatment (last treatment above 6 months).
  Interventions: Other: Additional biological samples
- Patients without cancer but aged above 70 years
  Interventions: Other: Additional biological samples
- Healthy person
  Interventions: Other: Additional biological samples

INTERVENTIONS:
Other: Additional biological samples — Peripheral Blood Mononuclear Cell (PBMC) and plasma will be collected

SUMMARY:
T-cell adaptive immunity is known to be required to sustain a long term immunoglobulin production and a long term memory against several infections. Previous results suggest a lack in the generation of T-cell responses against CoV-N, M and S proteins among cancer patients exposed to SARS-CoV-2 virus highlighting that cancer patients failed to mount a protective T-cell immunity. Given this context, our hypothesis is that COVID-19 vaccine candidates are not immunogenic in some cancer patients. Thus, the monitoring of CD4 and CD8 T-cell responses before and after vaccination might provide information related to the correlation between induction of CD4 T-cells (including helper follicular T-cells) by the vaccine and long-term IgG production (serological index). Additionally, the failure of COVID-19 vaccines in some patients should be monitor carefully in order to provide specific recommendations to avoid COVID-19 infections. The main objective is to assess humoral immune responses following COVID-19 vaccination in a population of cancer patients.

ELIGIBILITY:
*Inclusion Criteria:

* Male or female patients
* Age ≥ 18 years
* Not having developed a symptomatic form of COVID-19 within the last 3 months before inclusion
* Eligible to the vaccination against SARS-CoV-2
* Affiliation to French social security or receiving such a regime,
* Signed informed consent
* Ability to comply with the study protocol, in the Investigator's judgment

Cancer patients

* Patients under active anticancer treatment: in adjuvant or neoadjuvant setting or in first line of treatment in metastatic setting. Except for prostate cancer (until metastatic castration-resistant prostate cancer); and breast cancer hormonal receptor positive/HER2 negative (until apparition of hormonal resistance).
* Patients in follow-up (active treatment < 3 months).

Elderly:

Age ≥ 70 years old

Healthy person:

Age ≥ 18 years old and < 70 years old

*Exclusion Criteria:

* Patient under guardianship, guardianship or under the protection of justice
* Receipt of a live, attenuated vaccine within 4 weeks prior to the initiation of treatment or anticipation that such a live, attenuated vaccine will be required during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients vaccinated against COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2022-03-25 (Estimated); Study Completion 2023-03-25 (Estimated)

PRIMARY OUTCOMES:
Rate of virus-specific IgG at 3 months following COVID-19 vaccination measured in plasma to assess humoral immune responses | 2 years

SECONDARY OUTCOMES:
Rate of virus-specific IgG at 6 months following COVID-19 vaccination measured in plasma to assess humoral immune responses. | 2 years
Frequency of SARS-CoV-2 specific T-cell at 3 and 6 months following COVID-19 vaccination | 2 years
Magnitude of SARS-CoV-2 specific T-cell at 3 and 6 months following COVID-19 vaccination | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Marie KROEMER, Besançon, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gomez-Cadena A, Spehner L, Kroemer M, Khelil MB, Bouiller K, Verdeil G, Trabanelli S, Borg C, Loyon R, Jandus C. Severe COVID-19 patients exhibit an ILC2 NKG2D+ population in their impaired ILC compartment. Cell Mol Immunol. 2021 Feb;18(2):484-486. doi: 10.1038/s41423-020-00596-2. Epub 2020 Dec 14. No abstract available. PMID 33318627
- [Result] Kroemer M, Spehner L, Vettoretti L, Bouard A, Eberst G, Pili Floury S, Capellier G, Lepiller Q, Orillard E, Mansi L, Clairet AL, Westeel V, Limat S, Dubois M, Malinowski L, Bohard L, Borg C, Chirouze C, Bouiller K. COVID-19 patients display distinct SARS-CoV-2 specific T-cell responses according to disease severity. J Infect. 2021 Feb;82(2):282-327. doi: 10.1016/j.jinf.2020.08.036. Epub 2020 Aug 25. PMID 32853599
- [Derived] Spehner L, Orillard E, Falcoz A, Lepiller Q, Bouard A, Almotlak H, Kim S, Curtit E, Meynard G, Jary M, Nardin C, Asgarov K, Abdeljaoued S, Chartral U, Mougey V, Ben Khelil M, Lopez M, Loyon R, Vernerey D, Adotevi O, Borg C, Mansi L, Kroemer M. Predictive biomarkers and specific immune responses of COVID-19 mRNA vaccine in patients with cancer: prospective results from the CACOV-VAC trial. BMJ Oncol. 2023 Dec 14;2(1):e000054. doi: 10.1136/bmjonc-2023-000054. eCollection 2023. PMID 39886486